CLINICAL TRIAL: NCT02175368
Title: Clinical Evaluation of AdheSE One F Upgrade in Direct Filling Therapy
Brief Title: Adhese One F Upgrade in Direct Filling Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOFU 2012
Record Dates: First submitted 2014-06-20; First posted 2014-06-26 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Dental Adhesive
Keywords: total etch protocol; direct filling therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adhese One F Upgrade (Experimental): Adhese One F Upgrade (AOFU) is administered after phosphoric acid etching (etch-and-rinse protocol).
  Interventions: Device: Adhese One F Upgrade

INTERVENTIONS:
Device: Adhese One F Upgrade

SUMMARY:
Investigation on the clinical performance of a new dental adhesive when used in direct filling therapy after phosphoric acid etching.

Hypothesis: The new adhesive shows an acceptable clinical performance and allows a good filling quality.

ELIGIBILITY:
Inclusion Criteria:

* indication for class I or II filling
* max. 2 restorations per patient
* vital teeth
* sufficient language skills

Exclusion Criteria:

* dry working field cannot be established
* if the patient is known to be allergic to any of the materials' ingredients
* severe systemic diseases
* pregnancy
* non-vital or pulpitic teeth
* indication for indirect restoration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Peschke, Dr., Principal Investigator — Ivoclar Vivadent AG

RESULTS

PARTICIPANT FLOW:
Groups:
- Adhese One F Upgrade: Adhese One F Upgrade (AOFU) is administered after phosphoric acid etching (etch-and-rinse protocol).
  Adhese One F Upgrade
Period: Overall Study
Arm/Group | Adhese One F Upgrade
Started | 28
Completed | 27
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adhese One F Upgrade
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Liechtenstein | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success
Description: Clinical success is defined as no postoperative hypersensitivity and no loss of the restoration.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Adhese One F Upgrade
Number analyzed (Participants) | 28
Participants | 28

2. Secondary Outcome: Clinical Quality
Description: The clinical quality of the restorations will be evaluated according to semi-quantitative clinical evaluation (SQUACE) criteria and compared at all time points and at the end of the study.
  SQUACE is a published semi-quantitative method to evaluate the clinical success of dental restorations that is based on the commonly used USPHS criteria. The quality of the restoration is rated according to the SQUACE scale and classified as acceptable (patients with satisfactory clinical outcome) or not acceptable (patients with unsatisfactory clinical outcome).
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Adhese One F Upgrade
Number analyzed (Participants) | 28
Participants
  Patients with satisfactory clinical outcome | 28
  Patients with unsatisfactory clinical outcome | 0

ADVERSE EVENTS:
Arm/Group | Adhese One F Upgrade
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes